CLINICAL TRIAL: NCT02734017
Title: Impact of a Medication Review on Hospital Readmission: Study Protocol of a Randomized Controlled Trial
Brief Title: Impact of a Medication Review on Hospital Readmission: (ConcReHosp)
Acronym: ConcReHosp
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2015-20
Record Dates: First submitted 2016-03-23; First posted 2016-04-12 (Estimated); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Re-hospitalization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- standard course (Other): group not receiving medication review
  Interventions: Other: pharmacist-led standardized medication review
- pharmacist-led standardized medication review (Other): pharmacist-led standardized medication review including :
  * Medical and pharmaceutical admission medication reconciliation and treatment review
  * Medical and pharmaceutical medication reconciliation at discharge and treatment review
  * Medication Liaison Service
  Interventions: Other: pharmacist-led standardized medication review

INTERVENTIONS:
Other: pharmacist-led standardized medication review — the goal of this study is to assess the impact of the standardized medication review on the rate of readmissions and/or death at 30 days following initial hospitalization discharge.

SUMMARY:
The study is a randomized controlled clinical trial. A total 1400 hospitalized patients will be randomized in two groups:

1. group receiving a pharmacist-led standardized medication review (experimental group); and
2. group not receiving the medication review (control group).

The patients will be followed up at 30 days after initial hospitalization. Outcome measures include the number of readmissions; patient satisfaction, quality of medical admission prescription and number of consultation after initial hospitalization.

Discussion: A randomized controlled trial will provide the highest level of evidence on the impact of pharmacist-led standardized medication review on early hospital readmission for extreme age population.

DETAILED DESCRIPTION:
The impact of Medication Reconciliation on the early hospital readmission in the elderly is not clearly demonstrated. Moreover, the impact of medication reconciliation in the pediatric population is poorly studied.

In such context, it is important to demonstrate the effectiveness of the medication reconciliation as part of a standardized medication review process, in pediatric and in the elderly, on all cause readmissions in a large randomized control clinical trial. The standardized medication review process includes medication reconciliation, treatment review and medication liaison service.

The main objective of this study is to assess the impact of the standardized medication review on the rate of readmissions and/or death at 30 days following initial hospitalization discharge.

Methods/design: The study is a randomized controlled clinical trial. A total 1400 hospitalized patients will be randomized in two groups:

1. group receiving a pharmacist-led standardized medication review (experimental group); and
2. group not receiving the medication review (control group).

The patients will be followed up at 30 days after initial hospitalization. Outcome measures include the number of readmissions; patient satisfaction, quality of medical admission prescription and number of consultation after initial hospitalization.

Discussion: A randomized controlled trial will provide the highest level of evidence on the impact of pharmacist-led standardized medication review.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged under 18 or over 65 years
* Subject hospitalized in the multidisciplinary pediatric service or internal medicine ward, after emergency department visit at Timone hospital (Marseille, France) regardless of the reason for admission
* Subject with or without any comorbidity
* Living in France
* With national publicly-founded health insurance

Inclusion criteria for parents of minor child:

* Major subject and/or holder of parental authority of a hospitalized child, who fulfills the eligibility criteria mentioned above, in the multidisciplinary pediatric ward;
* Whatever the reason for hospitalization of the patient;

Inclusion criteria for the caregivers of patients older than 65 years:

* Major subject, designated by the patient or designating himself as the person most involved in the daily life of the patient;
* Whatever the reason for hospitalization of the patient;
* Whatever relationship or proximity to the study patient (family member, friend, neighbor);

Exclusion Criteria:

* Patients whose care requires regular re-hospitalization / programmed less than 30 days after discharge of initial hospitalization
* Vulnerable persons according to French law (pregnant women, adults under guardianship, persons deprived of liberty)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 470 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2019-01-02 (Actual); Study Completion 2019-03-23 (Actual)

PRIMARY OUTCOMES:
Rate of readmission | 30 days

SECONDARY OUTCOMES:
Satisfaction with Medicines Questionnaire (SatMed-Q®) | 30 days
  Patient satisfaction with regards to its drug treatment will be measured using the standardized questionnaire "Satisfaction with Medicines Questionnaire (SatMed-Q®)" validated in French
Medication errors on medical admission prescription | 24 hours
  Medical admission prescription will be assessed using the number of discrepancies and the number of medication errors,
Number of consultations post discharge | 30 days
  The number of consultations scheduled or not within 30 days' post-hospitalization will be studied. Consultations are defined as interviews with the attending physician, a specialist physician, nurse, therapeutic educator, and psychologist.

CONTACTS AND LOCATIONS:
Overall Officials: Urielle DESALBRES, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Hôpital de la Timone Assistance Publique Hôpitaux de Marseille, Marseille, France

REFERENCES:
- [Derived] Renaudin P, Baumstarck K, Daumas A, Esteve MA, Gayet S, Auquier P, Tsimaratos M, Villani P, Honore S. Impact of a pharmacist-led medication review on hospital readmission in a pediatric and elderly population: study protocol for a randomized open-label controlled trial. Trials. 2017 Feb 9;18(1):65. doi: 10.1186/s13063-017-1798-6. PMID 28183322